CLINICAL TRIAL: NCT04876508
Title: The Efficacy of Acupressure in Managing Opioid-induced Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Aydın University (Other)
Collaborators: Acibadem University (Other); Istanbul University (Other)
Responsible Party: Principal Investigator, DİLEK YILDIRIM, Assistant Professor, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OPIOID-INDUCED CONSTIPATION
Record Dates: First submitted 2021-05-01; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Opioid-induced Bowel Dysfunction; Constipation Drug Induced
Keywords: Acupressure; Constipation; Opioids-induced constipation; Complementary medicine
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure group (Experimental): Patients in the acupressure group will be given acupressure once a day for 7 consecutive days. Acupressure application will be applied by researchers who have been trained and certified on this subject. While the patients are in supine position, pressure will be applied to each acupressure point around the navel, respectively, Zhongwan (CV12), Guanyuan (CV4) and Tianshu (ST25) for 2 minutes for a total of 6 minutes.
  Interventions: Other: Accupressure
- Control group (No Intervention): No intervention will be applied

INTERVENTIONS:
Other: Accupressure — Patients in the experimental group will be given acupressure once a day for 7 consecutive days. Acupressure application will be applied by researchers who have been trained and certified on this subject. While the patients are in supine position, pressure will be applied to each acupressure point around the navel, respectively, Zhongwan (CV12), Guanyuan (CV4) and Tianshu (ST25) for 2 minutes for a total of 6 minutes.
  Arms: Acupressure group

SUMMARY:
In a randomized controlled study to evaluate the effect of acupressure application on opioid-related constipation, the Patient Identification Form, Defecation Diary, Visual Analog Scale and Constipation Quality of Life Scale will be applied after obtaining written informed consent from the patients. Patients in the experimental group will be given acupressure once a day for 7 consecutive days. Acupressure application will be applied by researchers who have been trained and certified on this subject. While the patients are in supine position, pressure will be applied to each acupressure point around the navel, respectively, Zhongwan (CV12), Guanyuan (CV4) and Tianshu (ST25) for 2 minutes for a total of 6 minutes. No attempt will be made to the control group. All patients will be followed for a total of 4 weeks and the Defecation Diary and Visual Comparison Scale will be applied weekly. 4. Constipation Quality of Life Scale will be applied again at the end of the week. The study was planned to examine the effect of acupressure on opioid-related constipation.

DETAILED DESCRIPTION:
Constipation symptom, which is very common in patients using opioids, affects the quality of life of the patients and may increase the severity of other symptoms. Pharmacological and non-pharmacological methods can be used in the management of opioid-associated constipation. One of the non-pharmacological approaches used is acupressure application. The effects of acupressure to increase bowel movements have been shown in studies. The study was planned to examine the effect of acupressure on opioid-related constipation. The goals that achieve this goal; To evaluate gastrointestinal functions in patients using opioid drugs, to examine and alleviate the effect of acupressure application on gastrointestinal functions (stool frequency, stool type, abdominal distension, abdominal pain, abdominal tenderness) in these patients, their quality of life (anxiety / anxiety states, physical, psychological discomfort) to evaluate and improve situations, satisfaction situations).

Study Population and Sample The research will be conducted in Istanbul University Istanbul Faculty of Medicine Hospital Algology Outpatient Clinic and Service. The universe of the study will consist of all patients followed in the Algology outpatient clinic and service. The sample of the study will consist of all patients who meet the inclusion criteria and who are willing to participate in the study. The patients enrolled in the study will be divided into intervention and control groups using the previously prepared randomization checklist.

Procedures In a randomized controlled study to evaluate the effect of acupressure application on opioid-related constipation, the Patient Identification Form, Defecation Diary, Visual Comparison Scale and Constipation Quality of Life Scale will be applied after obtaining written informed consent from the patients. Patients in the intervention group will be given acupressure once a day for 7 consecutive days. Acupressure application will be applied by researchers who have been trained and certified on this subject. While the patients are in supine position, pressure will be applied to each acupressure point around the navel, respectively, Zhongwan (CV12), Guanyuan (CV4) and Tianshu (ST25) for 2 minutes for a total of 6 minutes. No attempt will be made to the control group. All patients will be followed for a total of 4 weeks and the Defecation Diary and Visual Comparison Scale will be applied weekly.No intervention will be applied to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over who agreed to participate in the study,
* Cooperative and have no communication problem,
* Who have been on opioid therapy for at least 2 weeks,
* Can be fed orally,
* Constipation diagnosed by the physician,
* Patients whose constipation continues despite receiving laxative therapy for at least 1 week

Exclusion Criteria:

* Diagnosed with a known psychiatric illness (delirium, anxiety, panic attack, depression)
* Have thrombocytopenia (thrombocyte count <50,000 / μL),
* Have a gastrointestinal tumor,
* Having a history of abdominal hernia, bowel cancer and abdominal surgery,
* Having intraabdominal infection,
* Have irritable bowel syndrome and intestinal obstruction,
* Patients with inflammatory bowel disease will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient Information Form | Baseline
  The descriptive characteristics, age, gender, marital status, education status, diagnosis are included. It is 10 items in total.
Defecation diary- the amount of stool | patients will record their defecation status for 4 weeks each time they defecate.
  None (0) Less (+) (1) Medium (++) (2) It is scored as extra (+++) (3).
  As the score increases, constipation decreases. Includes a minimum of 0 and a maximum of 3 points.
Defecation diary - stool consistency | patients will record their defecation status for 4 weeks each time they defecate.
  Small, hard like marble (1 point) Bulky, hard (2 point) Normal (3 point) Soft (4 point) Aqueous (5 point)
  As the score increases, constipation decreases. Includes a minimum of 1 and a maximum of 5 points.
Defecation diary - straining during defecation | patients will record their defecation status for 4 weeks each time they defecate.
  Defecation without straining (1) Straining at the beginning of defecation (2) Straining in half defecation (3) Straining during all defecation (4)
  The higher the score, the higher the severity of constipation. Includes a minimum of 1 and a maximum of 4 points.
Defecation diary - feeling of incomplete emptying after defecation | patients will record their defecation status for 4 weeks each time they defecate.
  Present after defecation (1) None after defecation (0)
  The higher the score, the higher the severity of constipation. Includes a minimum of 0 and a maximum of 1 points.
Visual Analog Scale | this assessment on a daily basis, and a one-week total score was obtained for each item
  Pamuk et al. The form developed by (2003) includes 6 questions about the severity of the constipation symptoms. The Visual Analog Scale is a 10 cm horizontal line with 0 at one end and 10 at the other. The patient will be asked to mark the severity of each of the constipation symptoms on the horizontal line, giving a score between 0 and 10. The patients made this assessment daily, and by adding the scores, the total score average for one week for each item will be obtained. Minimum 0 Maximum 60 points are obtained from the scale. As the score increases, the severity of constipation increases.
Constipation Quality of Life Scale | Baseline and at the end of the fourth week
  It will be used in order to determine the effects of constipation related to opioid treatment on daily life and to measure the quality of life. The highest score that can be obtained from the scale is 140 and the lowest score is 28. It is thought that as the scores obtained from the scale increase, the quality of life is also negatively affected.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yildirim D, Kocatepe V, Talu GK. The efficacy of acupressure in managing opioid-induced constipation in patients with cancer: A single-blind randomized controlled trial. Support Care Cancer. 2022 Jun;30(6):5201-5210. doi: 10.1007/s00520-022-06947-1. Epub 2022 Mar 7. PMID 35257230